CLINICAL TRIAL: NCT00824993
Title: A Randomized, Controlled Study of Ibandronate for the Prevention of Bone Loss in Patients Who Have Received Allogeneic Bone Marrow Transplantation for Hematological Malignancies
Brief Title: Prevention of Osteoporosis in Bone Marrow Transplantation (BMT) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0960; NCI-2010-01024 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Hematological Malignancies
Keywords: Blood Cancer; Calcium; Vitamin D; Ibandronate; Boniva; Hematological Malignancies; Bone Marrow Transplantation; BMT; Osteoporosis; Bone Loss; Allogeneic Bone Marrow Transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Osteoporosis; Bone Diseases, Metabolic | interventions — Ibandronic Acid; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibandronate + Calcium + Vitamin D (Experimental): Ibandronate infusion of 3 mg by vein over 15 to 30 seconds for 4 doses at 3-6 weeks after transplant, and at Months 3, 6, and 9 after the transplant. Calcium 500 mg by mouth everyday for 12 months. Vitamin D 400 units by mouth 2 times a day for 12 months.
  Interventions: Drug: Ibandronate; Drug: Vitamin Supplements
- Calcium + Viatmin D (Experimental): Calcium 500 mg by mouth everyday for 12 months. Vitamin D 400 units by mouth 2 times a day for 12 months.
  Interventions: Drug: Vitamin Supplements

INTERVENTIONS:
Drug: Ibandronate — Infusion of 3 mg by vein over 15 to 30 seconds for 4 doses at 3-6 weeks after transplant, and at Months 3, 6, and 9 after the transplant.
  Other Names: Boniva
  Arms: Ibandronate + Calcium + Vitamin D
Drug: Vitamin Supplements — Calcium 500 mg by mouth everyday for 12 months
  Vitamin D 400 units by mouth 2 times a day for 12 months

SUMMARY:
The goal of this clinical research study is to see if ibandronate can help to slow the rate of bone loss that may occur in patients who have received a bone marrow transplant for blood cancer.

This study plans to address the following hypotheses:

1. The addition of Ibandronate initiated immediately after the transplantation will prevent bone loss in patients undergoing allogenic bone marrow transplantation (BMT) with underlying hematologic malignancies or hematologic disorders.
2. BMT patients who require prolonged steroid and other immunosuppressive treatment for Graft versus Host Diseases(GVHD) have a higher rate of bone loss, which can be prevented or attenuated by Ibandronate.

Specific objectives to test these hypotheses are:

1. Primary Objective:

   1. To prospectively compare the bone mineral density changes of lumbar spine, femoral neck and total hip between patients randomly assigned to ibandronate and control group over 12 months post bone marrow transplantation at the University of Texas MD Anderson Cancer Center.
2. Secondary Objectives:

   1. To measure and compare the accumulated level of steroid used in both treatment and control groups.
   2. To collect and compare the level of serum C-terminal telopeptide (CTX) in both treatment and control groups to monitor the bone turnover rate for the duration of the study.
   3. To conduct a cost-effectiveness analysis of participating patients for both outcomes on bone mineral density (measured data) and skeletal-related events (modeled data).
   4. To record incidence of bone fractures and the graft rate in both treatment and control groups.

DETAILED DESCRIPTION:
The Study Drug:

Ibandronate is designed to slow the rate of bone loss.

Screening Process:

Before you can receive the study drug, the study doctor will check the results of various tests that you recently had performed as part of standard care for the bone marrow transplant. These test results will help the doctor decide if you are eligible to take part in this study.

Study Groups:

If you are found to be eligible to take part in the study and you choose to take part, you will be randomly assigned (as in the toss of a coin) to 1 of 2 study groups. Group 1 (the "treatment" group) will receive ibandronate in addition to calcium and vitamin D supplements. Group 2 will only receive the calcium and vitamin D supplements. The chance of being in either group is equal.

Study Visits:

For both groups, you will be visited by a research team member during your hospital stay soon after the transplant (at Month Zero [0]), and during routine visits to your transplant doctor's office at Months 3, 6, and 9 after the transplant. At each of these study visits, you will be asked how you are feeling, as well as whether you have had any bone fractures (breakages).

At Months 0, 3, 6, and 9 after the transplant, blood (up to 1 tablespoon each time) will be drawn for routine tests for your transplant follow-up. As part of this same blood draw, an additional ½ tablespoon of blood will be drawn during each study visit (at Months 0, 3, 6, and 9). This blood will be tested for a "marker" in the bone that may help researchers predict who may respond to treatment.

If you are in the "treatment" group, you will receive a total of 4 ibandronate infusions by vein (over 15-30 seconds each time). These study drug infusions will take place in the hospital or at your routine visit to the transplant doctor's office at 3-6 weeks after the transplant, and at Months 3, 6, and 9 after the transplant.

At Month 6, all study participants will have a study-related (non-routine) bone density test (an x-ray) performed to check for bone loss. If the test results show that you have lost an abnormally large amount of bone mineral, you will be taken off study and also advised about treatment options.

Vitamin Supplements:

All study participants will receive a supply of calcium and vitamin D to take at home, for general bone health. These supplements should be taken by mouth, twice a day for 12 months. If you do not tolerate the supplements provided by the research study, you may take another brand of calcium/Vitamin D that you buy over-the-counter. The doses that you take each time (twice daily) should be 500 mg for calcium and 400 International Units (IU) for Vitamin D.

Cost Analysis:

Researchers on this study also want to look at how cost-effective the different procedures and treatments are on this study. To do this, they will use information from your patient records, pharmacy records, and other information of yours on M. D. Anderson databases. You will not be asked to actively participate in any interviews or procedures for these studies, but you should be aware that this research will take place while you are study.

End-of-Study Visit:

You will be visited by a research team member during your routine visit to your transplant doctor's office at Month 12 after the transplant. At this visit, you will be asked how you are feeling as well as whether you have had any bone fractures. Your doctor will check this by x-ray, if you do not have an outside x-ray film available. Blood (up to 1 tablespoon) will be drawn for routine tests. As part of this same blood draw, an additional ½ tablespoon of blood will be drawn to test for the same bone marker. You will have a routine bone density test (an x-ray) performed to check for bone loss. After these tests, your participation in this study will be over.

This is an investigational study. Ibandronate is commercially available and FDA approved for use in the prevention and treatment of bone loss in women who have been through menopause. However, its use in slowing the rate of bone loss in patients who have had a bone marrow transplant is considered experimental. For this purpose, the M. D. Anderson Institutional Review Board (IRB) has authorized the use of ibandronate for research only. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner.

Up to 200 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Patients with the diagnosis of hematologic malignancies or hematological disorders, who are immediately post- allogeneic bone marrow transplantation.
3. Female patients of childbearing potential (i.e. no hysterectomy, no loss of menses for 12 consecutive months), must be willing to use contraception.
4. Negative pregnancy test in premenopausal patients.
5. Patients with GVHD or infections can be entered only if they respond to treatment and become controlled.
6. Dental considerations: patients with negative dental screening for jaw osteonecrosis 0-3 months prior to their transplant and patients that do not have a plan for tooth extraction in the near future.

Exclusion Criteria:

1. Patients with documented relapsed malignancy or recurrence of the original hematological disorder after the transplant, uncontrolled acute GVHD, or uncontrolled infection.
2. Patients with hypocalcemia of less than 8.4 (corrected to account for the albumin level).
3. Patients with hypercalcemia >12.2, due to a cause not related to their hematological malignancy or hematological disorder (i.e. hyperparathyroidism, multiple myeloma).
4. Hypersensitivity to Ibandronate or other bisphosphonates.
5. Pre-existing osteoporosis, defined as a bone density T-score of -2.5 S.D. or less.
6. Renal insufficiency (calculated creatinine clearance < 30 ml/min).
7. Patients already on bisphosphonates (over the past two years), calcitonin, anabolic steroids, or daily oral fluoride supplement.
8. Myeloma patients who have previously been on bisphosphonates over the past two years and/or have active bone lesions.
9. If corrected calcium is above 10.3 and the immunoreactive parathyroid hormone (iPTH) is elevated or normal, the patient will be excluded from the study.
10. Patients with a 25-hydroxyvitamin D concentration <20 ng/ml and evidence of osteomalacia (low ionized calcium and elevated intact PTH).
11. Dental considerations: Patients with recent tooth extraction with signs of incomplete healing or significant infection will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-12-09 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Lu, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, randomized, placebo-controlled trial. Eligible patients were at least 18 years old and had undergone an allo-SCT for hematologic malignancy treatment within 45 days.
Pre-assignment Details: We screened 414 patients and 78 were enrolled.
Groups:
- Ibandronate: One 3 mg dose of ibandronate i.v. over 15 to 30 seconds at entry, 3, 6 and 9 months after allo-SCT, and elemental calcium 500 mg and vitamin D 800 IU per day for 12 months
- Control: Elemental calcium 500 mg and vitamin D 800 IU per day for 12 months
Period: Overall Study
Arm/Group | Ibandronate | Control
Started | 39 | 39
6 Month Follow up | 33 | 27
Completed | 25 | 22
Not Completed | 14 | 17
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Malignancy Relapse | 9 | 10
Not completed — Rapid Bone Loss | 0 | 1
Not completed — Non-Compliant | 2 | 1
Not completed — Insurance Issue | 2 | 1
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: All patient's enrolled in the study were analyzed (Intention To Treat)
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibandronate | Control | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 35 | 71
  >=65 years | 3 | 4 | 7
Age, Continuous [Median (Full Range); unit: years] | 55 [20 to 68] | 53 [20 to 70] | 54 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 36 | 39 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Bone Mineral Density From Baseline to 6 and 12 Months
Description: The primary outcome measure was the percentage change in BMD in the lumbar spine, femoral neck and total hip at 6 and 12 months (±4 weeks) after allo-SCT relative to baseline.
Time Frame: Baseline to 6 months and Baseline to 12 months
Population: We analyzed changes in BMD from baseline only for those who had follow up BMD evaluated at 6 and 12 months
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ibandronate | Control
Number analyzed (Participants) | 39 | 39
Percentage change
  % change baseline to 6m, LS: number analyzed (Participants) | 33 | 27
  % change baseline to 6m, LS | 0.06 (4.03) | -2.61 (4.2)
  % change baseline to 6m, FN: number analyzed (Participants) | 32 | 27
  % change baseline to 6m, FN | -3.63 (4.18) | -4.85 (5.37)
  % change baseline to 6m, TH: number analyzed (Participants) | 32 | 27
  % change baseline to 6m, TH | -2.73 (3.88) | -4.72 (4.32)
  % change baseline to 12m, LS: number analyzed (Participants) | 24 | 23
  % change baseline to 12m, LS | 1.27 (5.29) | -1.81 (4.49)
  % change baseline to 12m, FN: number analyzed (Participants) | 23 | 23
  % change baseline to 12m, FN | -4.29 (5.71) | -5.2 (5.25)
  % change baseline to 12, TH: number analyzed (Participants) | 23 | 23
  % change baseline to 12, TH | -4.85 (5.47) | -5.68 (5.15)

ADVERSE EVENTS:
Time Frame: Baseline to 12 months
Arm/Group | Ibandronate | Control
All-Cause Mortality (participants affected / at risk) | 1/39 | 3/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 21/39 | 24/39
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=39) | Control (N=39)
Infection - Other (Bacteremia) (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 6 | 4
Skin rash (Skin and subcutaneous tissue disorders) | 2 | 2
GI GVHD (Gastrointestinal disorders) | 0 | 4
Cystitis (Renal and urinary disorders) | 1 | 3
Fever (General disorders) | 1 | 2
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Other (Metabolism and nutrition disorders) | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-03-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT00824993/Prot_SAP_000.pdf